CLINICAL TRIAL: NCT00203320
Title: Etanercept for Alzheimer's-Type Memory Loss Pilot Study II
Brief Title: TNF-Alpha Inhibition for Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tobinick, Edward Lewis, M.D. (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10007
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2006-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: etanercept given by perispinal administration

SUMMARY:
It is widely believed that inflammation contributes to the pathogenesis of AD. TNF has been implicated in both AD and neurological inflammation. Anti-TNF therapy is therefore surmised to be of potential benefit for treating AD.

DETAILED DESCRIPTION:
Etanercept, a biologic anti-TNF fusion protein, will be administered weekly or biweekly by perispinal injection to a maximum of 30 study subjects for a period of one year with serial testing of cognition and function.

ELIGIBILITY:
Inclusion Criteria:

* NINCDS-ADRDA Criteria for Alzheimer's disease
* CT or MRI consistent with AD

Exclusion Criteria:

* active infection
* CHF
* demyelinating disease
* uncontrolled diabetes mellitus
* vascular dementia
* clinically significant neurologic disease other than AD
* Hachinski >4
* history of lymphoma
* TBC
* wbc<2500
* platelets<100,000
* HCT<30
* pregnancy
* premenopausal, fertile not on acceptable birth control
* change in neuroactive medication within 4 weeks of study initiation

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-04; Study Completion 2006-01

PRIMARY OUTCOMES:
ADAS-Cog
SIB
MMSE
ADCS-ADLsev

SECONDARY OUTCOMES:
Category fluency

CONTACTS AND LOCATIONS:
Overall Officials: Edward L. Tobinick, M.D., Principal Investigator — unaffiliated (Assistant Clinical Professor of Medicine, David Geffen School of Medicine at UCLA)
Locations (1):
- 100 UCLA Medical Plaza, Suites 205-210, Los Angeles, California, United States